CLINICAL TRIAL: NCT00480142
Title: Controlled Release of Oxycodone 10 mg In Pre-Medication For The Post Operative Analgesia In Elective Laparoscopic Bilateral Inguinal Hernia And Elective Laparoscopic Cholecystectomy : Prospective Double Blind, Randomized, Placebo-Controlled Study
Brief Title: Controlled Release of Oxycodone 10 mg In Pre-Medication For The Post Operative Analgesia In Elective Laparoscopic Bilateral Inguinal Hernia And Elective Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kmc070012CTIL
Record Dates: First submitted 2007-04-26; First posted 2007-05-30 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-05

CONDITIONS: Elective Laproscopic Bilateral Inguinal Hernia; Elective Laproscopic Cholecystectomy
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxycodone 10 mg

SUMMARY:
A Prospective Double Blind RCT: Controlled Release Oxycodone 10 mg On a 12 h Dosing Schedule Started With The Premedication ,Placebo Controlled Study,On Post Operative Analgesia Management in Laparoscopic Cholecystectomy and Laparoscopic Bilateral Inguinal Hernia (BIH).

CRO is indicated for the management of moderate to severe pain when a continuous,around the clock analgesic is needed for an extended period of time.Its safety and efficacy in the first 12-24 hours post operative has not been established.

ELIGIBILITY:
Inclusion Criteria:

* Local ethic committee approval
* Written informed consent
* ASA physical status I-III, scheduled for elective laparoscopic cholecystectomy and elective laparoscopic BIH

Exclusion Criteria:

* Difficulty in communication
* Allergy to oxycodone and/or morphine
* Allergy to local anesthetic
* History of alcohol and substance abuse
* Treated depression
* Chronic use of opioid or tramadol or NSAIDS
* Pregnancy
* Obstructive sleep apnea
* Anticipated fiber optic intubation
* Severe hepatic or renal impairment
* Weight <50 kg or > 100 kg
* Conversion to laparotomy
* Patient extubated in PACU.
* Any prior abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Study Completion 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: patricia grosman, MD, Principal Investigator — Israel: Kaplan Hospital, Clalit Health Service; Eli Mavor, MD, Study Chair — Israel:Clalit Health Service; oscar liphshitz, MD, Study Director — Isreal: Kaplan: Clalit Health Service; Bella Almog, R.N MA, Study Director — Israel: Kaplan: Clalit Health Service